CLINICAL TRIAL: NCT00122122
Title: Randomized Controlled Trial of Enhanced Pharmacy Care in Older Veteran Outpatients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAF 98-152
Record Dates: First submitted 2005-07-18; First posted 2005-07-21 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Geriatrics; Drug Therapy; Poly Pharmacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Enhanced Pharmacy Care

INTERVENTIONS:
Behavioral: Enhanced Pharmacy Care

SUMMARY:
Complications resulting from medications, or adverse drug events (ADEs), are prevalent and are a major source of excess morbidity and costs. ADEs are particularly problematic in older patients because of their higher burden of comorbidity and diminished physiologic reserve. In addition, older patients are more likely to be exposed to polypharmacy, a major risk factor for ADEs. While ADEs may be idiosyncratic, many result from medical errors and inadequate systems for ensuring the safe and effective use of medications.

The goal of the proposed study is to test the efficacy of a potentially potent intervention to improve the use of medications in older outpatients enrolled in VA primary care clinics. The intervention-Enhanced Pharmacy Care-involves a formal, multi-dimensional evaluation of patients� medication regimens by a trained clinical pharmacist and board-certified geriatrician.

DETAILED DESCRIPTION:
Background:

Complications resulting from medications, or adverse drug events (ADEs), are prevalent and are a major source of excess morbidity and costs. ADEs are particularly problematic in older patients because of their higher burden of comorbidity and diminished physiologic reserve. In addition, older patients are more likely to be exposed to polypharmacy, a major risk factor for ADEs. While ADEs may be idiosyncratic, many result from medical errors and inadequate systems for ensuring the safe and effective use of medications.

The goal of the proposed study is to test the efficacy of a potentially potent intervention to improve the use of medications in older outpatients enrolled in VA primary care clinics. The intervention-Enhanced Pharmacy Care-involves a formal, multi-dimensional evaluation of patients� medication regimens by a trained clinical pharmacist and board-certified geriatrician.

Objectives:

The study has the following six aims: 1) Compare changes in prescribing practices-as measured by medication appropriateness, number of medications, and cost of prescribed medications-between baseline and follow-up in patients randomized to Enhanced Pharmacy Care and patients randomized to usual care; 2) Compare other medication-based endpoints in the two groups, including the occurrence of potential ADEs, medication compliance, and patient knowledge of medications; 3) Compare changes in health-related-quality-of-life in the two groups; 4) Compare patient perceptions of the quality of VA outpatient care in the two groups; 5) Compare health care utilization during the one-year study period in the two groups; and 6) Examine attitudes of primary care providers (PCPs) about the intervention.

Methods:

Patients were eligible for the trial if they were 65 years and older and receiving prescriptions for > 5 medications in a VA primary care clinic. Patients were randomized to usual care or to the intervention, which included a structured medication history and medical records review. For intervention patients, therapeutic recommendations were developed and presented to primary care providers. Baseline and 3-month measures were obtained and change was assessed by analysis of covariance.

Status:

493 patients have been enrolled in the trial and 12-month follow-up has been completed on over 95% of patients. Preliminary results have been evaluated and abstracts have been submitted to national meetings, including the 2004 VA HSR&D and 2004 SGIM Annual Meetings where it will be presented as an oral presentation. We are completing all the data cleaning and will be performing final analyses on the data, with manuscript preparation. Final outcome assessment using the Medication Appropriateness Index is in the final stage.

ELIGIBILITY:
Inclusion Criteria:

Patients enrolled in VA primary care clinics who are 65 years and older and who are receiving prescriptions for 5 or more scheduled medications.

Exclusion Criteria:

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 600 (Estimated)
Dates: Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary E. Rosenthal, MD, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (1):
- Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa, United States

REFERENCES:
- [Result] Steinman MA, Rosenthal GE, Landefeld CS, Bertenthal D, Kaboli PJ. Agreement between drugs-to-avoid criteria and expert assessments of problematic prescribing. Arch Intern Med. 2009 Jul 27;169(14):1326-32. doi: 10.1001/archinternmed.2009.206. PMID 19636035
- [Result] Steinman MA, Rosenthal GE, Landefeld CS, Bertenthal D, Sen S, Kaboli PJ. Conflicts and concordance between measures of medication prescribing quality. Med Care. 2007 Jan;45(1):95-9. doi: 10.1097/01.mlr.0000241111.11991.62. PMID 17279026